CLINICAL TRIAL: NCT07171177
Title: Disability and Pain in Men and Women With Chronic Low Back Pain and Pronated Foot Treated With Custom-made Foot Orthoses
Brief Title: Disability and Pain in Chronic Low Back Pain and Pronated Foot Treated
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, MANUEL PABON CARRASCO, Principal Investigator, Assistant Professor, Faculty of Nursing, Physiotherapy and Podiatry, University of Seville, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: USev-Foot 2
Record Dates: First submitted 2021-04-26; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2021-04

CONDITIONS: Low Back Pain; Foot Orthoses; Pronation
MeSH Terms: conditions — Low Back Pain | interventions — Foot Orthoses

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Custom-made plantar orthosis (3 mm polyurethane foam + 3 mm polypropylene) (Experimental): Individually manufactured plantar orthosis, moulded to each patient's pronated foot using 3 mm polyurethane foam laminated with 3 mm polypropylene, designed to control excessive pronation and thus potentially alleviate non-specific chronic low back pain.
  Interventions: Device: Foot Orthoses
- Arm/Group Title: Placebo Comparator: Flat insole (placebo orthosis) (3 mm polyurethane foam) (Placebo Comparator): Flat insole made of 3 mm polyurethane foam without corrective elements, used as a placebo comparator to the custom-made orthosis in the management of non-specific chronic low back pain.
  Interventions: Device: Foot Orthoses

INTERVENTIONS:
Device: Foot Orthoses — To compare the use of handmade plantar orthoses versus the use of splints in the management of low back pain.

SUMMARY:
Purpose: excessive foot pronation has been reported as being related to chronic low back symptoms. Compensating custom-made foot orthotics treatment has not been entirely explored as an effective therapy for chronic low back pain (CLBP). This study aims to observe the effects of custom made foot orthoses, in subjects with foot pronation suffering from CLBP.

ELIGIBILITY:
Inclusion Criteria:

* Women and men adults up to 65 years old,
* presence of Chronic Low Back Pain
* Foot Posture Index pronated in one or both feet (henceforth, FPI) ≥ +6

Exclusion Criteria:

* Serious illness.
* Current participation in another research study.
* Pregnancy.
* Previous back or foot surgery
* Current treatment of a foot or back pathology
* Leg length discrepancy > 5 mm

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Change in disability due to low back pain measured by the Roland-Morris Disability Questionnaire (RMDQ) | Baseline and 4 weeks after intervention
  The RMDQ is a 24-item self-reported questionnaire designed to assess physical disability due to low back pain. Scores range from 0 to 24, with higher scores indicating greater disability.

SECONDARY OUTCOMES:
Change in pain intensity measured by the Numerical Rating Scale (NRS, 0-10) | Baseline and 4 weeks
  The NRS is a 0-10 scale where 0 = no pain and 10 = worst imaginable pain.
Change in foot posture measured by the Foot Posture Index (FPI) | Baseline and 4 weeks
  The FPI is a 6-item clinical tool for quantifying foot posture. Total scores range from -12 (highly supinated) to +12 (highly pronated).

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Sevilla, Seville, sevilla, Spain

IPD SHARING:
Plan to Share IPD: Undecided